CLINICAL TRIAL: NCT05666024
Title: Clinical Study on the Effect of Labor Analgesia on the Postpartum Recovery Outcome of Chinese Parturients
Brief Title: A Clinical Study on the Effect of Labor Analgesia on the Postpartum Recovery Outcome of Chinese Parturients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang，MD, Clinical Professor, Huazhong University of Science and Technology
Other Study IDs: Labor analgesia
Record Dates: First submitted 2022-12-02; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Analgesia; Labor Analgesia
Keywords: Labor analgesia; Chinese parturients; Postpartum recovery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parturients: Maternity about to give birth

INTERVENTIONS:
Other:  — Prospective observational study

SUMMARY:
Background:

The parturient will experience extreme pain during delivery. Effective labor analgesia will bring better delivery experience to the parturient, while the adverse experience during delivery may bring many adverse effects to the parturient, including postpartum depression, insomnia, and even suicide. Postpartum depression, which has a high incidence, is one of the most common diseases that affect the quality of life of pregnant women during the perinatal period. Postpartum depression even leads to maternal suicide, which is the main cause of maternal death in the first year after childbirth. At the same time, postpartum depression seriously affects the relationship between mother and baby, which significantly increases the risk of long-term psychological sequelae of their children. Its incidence in Europe and America is about 10%, while in China it even reaches 15.7-39.8%. In addition, these factors may also affect maternal breast milk and adversely affect the psychological and behavioral development of infants. Many studies report that effective analgesia can reduce the incidence of postpartum depression in the process of natural delivery, which indicates that labor analgesia is one of the effective measures to reduce postpartum depression. However, the sample size of these studies is relatively small, and they usually focus on the psychological impact on the mothers themselves, and the focus time is only 6-8 weeks after the operation. However, there is still a lack of large sample multicenter studies on the long-term outcome of postpartum mothers and newborns (including the impact of breast feeding and neonatal neurointellectual development).

Objective:

1. The subjects were included and comprehensive perinatal data were collected. On this basis, the database of maternal and neonatal prognosis for labor analgesia was established;
2. Different data analysis methods were used to analyze the differences of maternal and neonatal outcomes to provide evidence based medical evidence for the current situation of labor analgesia and the optimization of labor analgesia mode.

DETAILED DESCRIPTION:
Based on the principle of Real World Study (RWS), this study is intended to conduct a prospective observational study through long-term comprehensive outcome follow-up of a large sample of multiple centers, and then, based on different studies, conduct a synchronous survey by gathering comprehensive attention on outcome indicators, and use machine learning, regression analysis, propensity matching and other analysis methods for data analysis, Finally, independent analysis based on different sub research topics combined with big data analysis will provide effective evidence-based medical evidence for the optimization of current labor analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 20 ≤ age ≤ 45;
* ASA I ～ III;
* Willing to participate in this study and sign the informed consent form.

Exclusion Criteria:

* Take other trial drugs or participate in other clinical trials 3 months before inclusion in the study;
* Unable to cooperate with the research for any reason.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parturients
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Data collection and database establishment | 2024
  The subjects were included and comprehensive perinatal data were collected. On this basis, the prognostic database of parturients with labor analgesia and neonates was established

SECONDARY OUTCOMES:
data analysis | 2024
  Different data analysis methods are used to analyze the differences of maternal and neonatal outcomes, so as to provide evidence-based medical evidence for the current situation of labor analgesia and the optimization of labor analgesia mode.

CONTACTS AND LOCATIONS:
Overall Officials: Xianwei Zhang, Doctor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pollard K. MBRRACE-UK Report launch December 2016. Pract Midwife. 2017 Feb;20(2):30-2. PMID 30462430
- [Background] Pearson RM, Evans J, Kounali D, Lewis G, Heron J, Ramchandani PG, O'Connor TG, Stein A. Maternal depression during pregnancy and the postnatal period: risks and possible mechanisms for offspring depression at age 18 years. JAMA Psychiatry. 2013 Dec;70(12):1312-9. doi: 10.1001/jamapsychiatry.2013.2163. PMID 24108418
- [Background] Munk-Olsen T, Laursen TM, Pedersen CB, Mors O, Mortensen PB. New parents and mental disorders: a population-based register study. JAMA. 2006 Dec 6;296(21):2582-9. doi: 10.1001/jama.296.21.2582. PMID 17148723
- [Background] Howard LM, Molyneaux E, Dennis CL, Rochat T, Stein A, Milgrom J. Non-psychotic mental disorders in the perinatal period. Lancet. 2014 Nov 15;384(9956):1775-88. doi: 10.1016/S0140-6736(14)61276-9. Epub 2014 Nov 14. PMID 25455248
- [Background] Siu BW, Leung SS, Ip P, Hung SF, O'Hara MW. Antenatal risk factors for postnatal depression: a prospective study of Chinese women at maternal and child health centres. BMC Psychiatry. 2012 Mar 22;12:22. doi: 10.1186/1471-244X-12-22. PMID 22436053
- [Background] Wang SY, Jiang XY, Jan WC, Chen CH. A comparative study of postnatal depression and its predictors in Taiwan and mainland China. Am J Obstet Gynecol. 2003 Nov;189(5):1407-12. doi: 10.1067/s0002-9378(03)00673-2. PMID 14634578
- [Background] Goldbort J. Transcultural analysis of postpartum depression. MCN Am J Matern Child Nurs. 2006 Mar-Apr;31(2):121-6. doi: 10.1097/00005721-200603000-00012. PMID 16523038
- [Background] Lim G, Facco FL, Nathan N, Waters JH, Wong CA, Eltzschig HK. A Review of the Impact of Obstetric Anesthesia on Maternal and Neonatal Outcomes. Anesthesiology. 2018 Jul;129(1):192-215. doi: 10.1097/ALN.0000000000002182. PMID 29561267
- [Background] Ding T, Wang DX, Qu Y, Chen Q, Zhu SN. Epidural labor analgesia is associated with a decreased risk of postpartum depression: a prospective cohort study. Anesth Analg. 2014 Aug;119(2):383-392. doi: 10.1213/ANE.0000000000000107. PMID 24797120
- [Background] Lim G, Farrell LM, Facco FL, Gold MS, Wasan AD. Labor Analgesia as a Predictor for Reduced Postpartum Depression Scores: A Retrospective Observational Study. Anesth Analg. 2018 May;126(5):1598-1605. doi: 10.1213/ANE.0000000000002720. PMID 29239949
- [Result] Stewart DE, Vigod S. Postpartum Depression. N Engl J Med. 2016 Dec 1;375(22):2177-2186. doi: 10.1056/NEJMcp1607649. No abstract available. PMID 27959754